CLINICAL TRIAL: NCT06449690
Title: Interest of Animal-assisted Therapy With Dogs in the Treatment of Depression: a Randomized Controlled Trial
Brief Title: Interest of Animal-assisted Therapy With Dogs in the Treatment of Depression
Acronym: DATID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Bon Sauveur De La Manche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FBSM-001; N° ID-RCB : 2024-A00645-42 (Other: ANSM (France))
Record Dates: First submitted 2024-05-30; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Depression
Keywords: Depression; Dog-assisted therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dog-assisted therapy (Experimental): Patients in the "dog-assisted therapy" arm will participate in two group sessions (groups of 3 to 7 participants) of canine-assisted therapy, supervised by a healthcare professional certified in animal-assisted therapy alongside a psychiatric caregiver, for 30 minutes each week over 6 weeks.
  Interventions: Procedure: Dog-assisted therapy
- Occupational activities (Active Comparator): Patients in the "occupational activities" arm will participate in two group sessions (groups of 3 to 7 participants) of occupational activities, supervised by a healthcare professional experienced in group occupational activities alongside a psychiatric caregiver, for 30 minutes each week over 6 weeks.
  Interventions: Procedure: Occupational activities

INTERVENTIONS:
Procedure: Dog-assisted therapy — Dog-assisted therapy consists of the search for positive interactions resulting from the intentional human-animal relationship in the educational, therapeutic or social fields, practices as they are conducted in educational and medico-social institutions for example.
  Arms: Dog-assisted therapy
Procedure: Occupational activities — Occupational activities consist of origami, relaxation, sports or board games sessions.
  Arms: Occupational activities

SUMMARY:
This study is a randomized controlled trial (comparing "occupational activities" versus "dog-assisted therapy" arms) investigating the effectiveness of animal-assisted therapy with dogs in small groups of participants with depression. Patients in the "dog-assisted therapy" arm will participate in two group sessions (groups of 3 to 7 participants) of canine-assisted therapy, supervised by a healthcare professional certified in animal-assisted therapy alongside a psychiatric caregiver, for 30 minutes each week over 6 weeks. Patients in the "occupational activities" arm will participate in two group sessions (groups of 3 to 7 participants) of occupational activities, supervised by a healthcare professional experienced in group occupational activities alongside a psychiatric caregiver, for 30 minutes each week over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65
* Patient affiliated with a social security scheme
* Patient hospitalized under voluntary psychiatric care
* Diagnosis of depression according to DSM-5-TR criteria
* QIDS-C16 score ≥11 at screening
* QIDS-SR16 score ≥11 at screening and inclusion

Exclusion Criteria:

* Severe comorbid psychiatric disorder
* Imminent risk of suicidal behavior
* Unstable comorbid somatic condition
* Vulnerable patients (under guardianship, curatorship, or judicial protection)
* Known fear of dogs
* Known allergy to dog fur

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the 17-item Hamilton Depression Rating Scale (HDRS) score from baseline to 6 weeks. | Baseline and week 6
  The 17-item Hamilton Depression Rating Scale (HDRS) is a validated scale for depression assessment, its score is rated between 0 and 52 and a higher score means a more depressed state

SECONDARY OUTCOMES:
Evolution of the 17-item Hamilton scale score between 0 and 3 weeks. | Baseline and week 3
  The 17-item Hamilton Depression Rating Scale (HDRS) is a validated scale for depression assessment, its score is rated between 0 and 52 and a higher score means a more depressed state
Evolution of the quality of life scale score (WHOQOL-BREF) at 3 and 6 weeks, compared to the initial score at W0. | Baseline and weeks 3 and 6
  The World Health Organization Quality Of Life (WHOQOL) WHOQOL-BREF scale is a validated scale for the measurement of quality of life, its score is rated between 0 and 100 and a higher score means better quality of life
Evaluation of the number of adverse events and serious adverse events related to the therapy under study. | From baseline up to 6 weeks
  The number of AEs will be used to assess the safety of the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy MADIGAND, MD, Principal Investigator — Fondation Bon Sauveur De La Manche

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bousman CA, Arandjelovic K, Mancuso SG, Eyre HA, Dunlop BW. Pharmacogenetic tests and depressive symptom remission: a meta-analysis of randomized controlled trials. Pharmacogenomics. 2019 Jan;20(1):37-47. doi: 10.2217/pgs-2018-0142. Epub 2018 Dec 6. PMID 30520364
- [Background] Lundqvist M, Carlsson P, Sjodahl R, Theodorsson E, Levin LA. Patient benefit of dog-assisted interventions in health care: a systematic review. BMC Complement Altern Med. 2017 Jul 10;17(1):358. doi: 10.1186/s12906-017-1844-7. PMID 28693538
- [Background] Richerson JT, Wagner TH. Service Dogs for Veterans With PTSD. Psychiatr Serv. 2023 Jun 1;74(6):668-669. doi: 10.1176/appi.ps.20230164. No abstract available. PMID 37259586
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942